CLINICAL TRIAL: NCT05239962
Title: Evaluation of Reliability and Validity of Urdu Version of Spine Functional Index
Brief Title: A Reliability And Validity Study Of The Urdu Version Of Spine Functional Index.
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0289
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Spinal Deformity
Keywords: Spine Functional Index; Spinal Disorders; Cultural adaptation; Validity; Urdu Version; Reliability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Aim of the study is to translate Spine Functional Index scale into Urdu Language and to investigate the validity and reliability in Pakistan with the populace of Spinal disorders. Also checks its co-relation with Neck disability Index and Roland-Morris Disability Questionnaire.

DETAILED DESCRIPTION:
As per the previous recommendations, the Spine Functional Index will be interpreted in urdu language and adapted culturally. Participants will be selected by the convenience sampling technique based on pre-defined inclusion and exclusion criteria from a total of 220 participants with spinal Disorders. To test the reliability of Urdu Version Of Spine Functional Index, Neck Disability Index and Roland-Morris Disability Questionnaire in the inter and intra-observer environment, two observers and an interim interval of 45 minutes between the first and second application fill out a questionnaire on the same day for the inter-observer assessment. Observer-1 for the intra-observer evaluation will conduct a third evaluation after 7 days. Using Statistical Package of Social Sciences version 24, data is entered and analyzed. Cronbach Alpha Value is used to analyze center consistency. The intraclass correlation coefficient is used to assess the reliability of the test-retest. For content validity, criteria validity and responsiveness, the Urdu Version Of Spine Functional Index was assessed.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for participation in this study were at least 18 years of age.
* The patient must be diagnosed with musculoskeletal disorder of the spine.
* The patient can be chronic and sub-acute and acute.
* The patient can be referred by a physician or physical therapist.

Exclusion Criteria:

* Lack of reading Urdu or reply to the survey questions were the criteria for exclusion.
* Infectious diseases and patient without spinal disorders were excluded.
* The patients with late surgery or systemic sickness which effects spine was excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be of Spinal cord disorders like. Lumbar or thoracic or Cervical or Multiple Areas pain
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Spine Functional Index | 1st day
  Spine Functional Index is a single page of 25 items with a three-point respond option. The score of 25 items is summed and this score is then multiplied by four and deducted from 100 (0 % score = max disability or functional loss and 100 % score = no impairments or normal).
Roland-Morris Questionnaire | 1st day
  Roland-Morris Questionnaire is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale.
Neck Disability Index | 1st day
  Neck Disability Index contains total 50 scores. 5 marks for each statement. If the response is missing then the score will not be conducted or included in total marks.
Oswestry Low Back Pain Index | 1st day
  Oswestry Low Back Pain Index is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No